## **Statistical Analysis Plan**

**Identifier:** NCT02414607

Study Title: Effect of Elderberry Juice on Cognition and Inflammation in Patients With Mild

Cognitive Impairment

## Baseline demographics and clinical characteristics

Group differences between Elderberry and Placebo control were evaluated using independent sample t-tests for continuous variables and chi-square analyses for categorical variables.

## Cognitive Measures

For each outcome variable, fixed effects of group (Elderberry, Placebo control), time (baseline, 3-month follow-up; baseline, 6-month follow-up) and the group by time interaction will be tested using Multilevel Modeling (MLM) analyses in SPSS (version 27), using a first-order Autoregressive covariance structure (AR1) and restricted maximum likelihood estimation. Given the preliminary nature of the study, pairwise comparisons between groups and within groups over time will be examined for both significant effects (alpha  $\leq$  .05) and trends (alpha < .10).